CLINICAL TRIAL: NCT00675922
Title: Comparing the Use of Sulfamylon 5%, Dakins 0.025%, Cerium, Silver Nitrate 5% and/or Other Topical Antimicrobial Products for the Treatment of Excised and/or Grafted Burn Wounds
Brief Title: Study of the Treatment of Burn Wounds With Antimicrobial Topical Soaks
Acronym: Soaks
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Data inconclusive.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95-096
Record Dates: First submitted 2007-12-26; First posted 2008-05-12 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Burn
Keywords: Burn; Wounds; Wound infection; Topical antimicrobials; Cerium; Dakins; Sulfamylon Soaks; Silver Nitrate
MeSH Terms: conditions — Burns; Wounds and Injuries; Wound Infection | interventions — Mafenide; Silver Nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sulfamylon 5% and Silver Nitrate Soaks (Experimental): Application of Sulfamylon 5% Solution and Silver Nitrate soaked dressings to two different burned area. Sites were then monitored for infections during hospitalization.
  Interventions: Drug: Sulfamylon 5% and Silver Nitrate Soaks

INTERVENTIONS:
Drug: Sulfamylon 5% and Silver Nitrate Soaks — Application of Sulfamylon and Silver Nitrate Solution to burn wound daily
  Other Names: Sulfamylon; Silver Nitrate

SUMMARY:
Determine effectiveness of various antimicrobial solutions on burn wounds (infections, wound healing, length of hospital stay).

DETAILED DESCRIPTION:
Patients were treated with both Sulfamylon soaks and Silver nitrate soaks on different burn areas. These two areas were then compared for incidence (percentage) of infections.

ELIGIBILITY:
Inclusion Criteria:

* Burn Injury requiring excisional therapy
* Hospitalization required until wounds are closed

Exclusion Criteria:

* Known hypersensitivity to products
* Outpatient treatment for burn injury

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 1995-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to Burn ICU with acute burn injury were eligible for recruitment
Pre-assignment Details: Patients consented were randomized to one or two of the treatment medications.
Groups:
- Sulfamylon Solution 5% and Silver Nitrate Soaks: Application of Sulfamylon 5% and Silver Nitrate Solution soaked dressings to a burned area
Period: Overall Study
Arm/Group | Sulfamylon Solution 5% and Silver Nitrate Soaks
Started | 98
Completed | 98
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sulfamylon vs Silver Nitrate Solution: Application of Sulfamylon 5% and Silver Nitrate Solution soaked dressings to a burned area
Arm/Group | Sulfamylon vs Silver Nitrate Solution
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 66

OUTCOME MEASURES:

1. Primary Outcome: Infection Rate
Description: Percent of infections following antimicrobial topical treatment with Sulfamylon vs Silver Nitrate Soaks.
Time Frame: Acute hospitalization following burn injury: admission to discharge (1-20 weeks)
Population: Percent of sites treated with sulfamylon of Silver Nitrate soaks that developed infections
Measure: Number; unit: percentage of participants
Groups:
- Percent Infections:Sulfamylon Site: Percent of sites that developed infections with Sulfamylon soaks
- Percent Infections: Silver Nitrate Site: Percent of sites that developed infections with Silver Nitrate soaks
Arm/Group | Percent Infections:Sulfamylon Site | Percent Infections: Silver Nitrate Site
Number analyzed (Participants) | 98 | 98
percentage of participants | 72 (.05) | 74

2. Secondary Outcome: Length of Hospital Stay With Various Antimicrobial Solutions for Burn Patients
Description: At the request of the study site, this study has been closed. Access to study-related data is unavailable, and the PI is no longer at the institution. Hence, we are unable to submit the results data for this outcome. Although peer-reviewed articles have been located that reference NCT00675922 it is not clear and verifiable (without access to the actual study-related data) what the results for this outcome.
Time Frame: Admission to burn unit to discharge
Population: At the request of the study site, this study has been closed. Access to study-related data is unavailable, and the PI is no longer at the institution. Hence, we are unable to submit the results data for this outcome. Although peer-reviewed articles have been located that reference NCT00675922 it is not clear and verifiable (without access to the actual study-related data) what the results for this outcome.
Arm/Group | Percent Infections:Sulfamylon Site | Percent Infections: Silver Nitrate Site
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1995-2008
Groups:
- Sulfamylon Soaks, Silver Nitrate Soaks: Patients receive both treatments and each treated site is compared.
Arm/Group | Sulfamylon Soaks, Silver Nitrate Soaks
Serious Adverse Events (participants affected / at risk) | 9/98
Other Adverse Events (participants affected / at risk) | 2/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulfamylon Soaks, Silver Nitrate Soaks (N=98)
Invasive infection, MOF, death (Infections and infestations) | 1 (1) — 2001: 74% burn admitted with invasive infection, developed multi organ failure and expired. PI opinion is Adverse Event is unlikely related to study.
ischemia of leg (Vascular disorders) | 1 (1) — 2001: 80% burn patient, during Arterial IV line placement for surgery, right leg became ischemic. Anticoagulants given. Patient discharged without complications. PI opinion is Adverse Event is not related to study.
renal failure, death (Renal and urinary disorders) | 1 (1) — 2001: 90% burn admitted with renal failure. After patient was 95% grafted and healed, renal failure worsened and patient expired. PI opinion is Adverse Event unlikely related to study.
Patient aspiration and death (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 2001: 62% burn after discharge, patient aspirated during the night Advanced Cardiac Life Support provided, patient expired. PI opinion is Adverse Event not related to study.
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 2001: 70% burn patient, pneumothorax occured during subclavian IV line placement for surgery. PI opinion is Adverse Event is not related to study.
hypoglycemia (Endocrine disorders) | 2 (2) — 2001: 70% burn patient blood sugar decreased to 30 while on insulin drip. 2001: 70% burn patient blood glucose decreased to 35 while on insulin drip. PI opinion, Neither Adverse Event is related to study.
Sepsis, multi organ failure and death (Infections and infestations) | 1 (1) — 2001: 85% burn admitted with invasive infections became septic, developed renal failure then multi organ failure. Patient removed from respiratory support and expired. PI opinion, Adverse Event is possibly related to study.
chest tube fell out (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 2001: 70% burn, chest tube fell out while patient was being moved. PI opinion, Adverse Event not related to study.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulfamylon Soaks, Silver Nitrate Soaks (N=98)
skin, opened wound (Skin and subcutaneous tissue disorders) | 1 (1) — 42% burn, patient fell and opened a wound in groin area. PI opinion, Adverse Event not related to study.
open wound (Skin and subcutaneous tissue disorders) | 1 (1) — 2003: 42% burn patient scratched biopsy site that had been sutured shut, opening a wound. PI opinion, Adverse Event not related to study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No